CLINICAL TRIAL: NCT06933017
Title: Feasibility Study of the Augmented Two-Day 6-Minute Incremental Step Test and Causal Exploration Through a Directed Acyclic Graph and Structural Equation Model for Post-Exertional Symptom Exacerbations in Long COVID Patients
Brief Title: Feasibility of an Augmented Two-Day Step Test and Causal Modeling for Post-Exertional Symptom Exacerbation in Post Covid-19 Syndrome
Acronym: REVEAL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitair Ziekenhuis Brussel (Other)
Collaborators: Vrije Universiteit Brussel, Jette, Belgium (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Device Feasibility
Other Study IDs: 2024-EDW-REVEAL; G075423N (Other Grant/Funding Number: Fonds Wetenschappelijk Onderzoek)
Record Dates: First submitted 2025-04-03; First posted 2025-04-17 (Actual); Last update posted 2025-07-08 (Actual); Status verified 2025-02

CONDITIONS: Long COVID
Keywords: long covid; PEM; Post-Exertional Malaise; CPET; 6MIST; Fatigue
MeSH Terms: conditions — Post-Acute COVID-19 Syndrome; Fatigue

STUDY DESIGN:
Intervention Model Description: Feasibility study in a cross-over model. The investigators calculated 40% drop out because this protocol presents considerable challenges for participants to complete.
Masking Description: Statistician
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Two day 6-Minute Incremental Step Test (6 MIST) (Experimental): The 6-Minute Incremental Step Test (6MIST) is an incremental pace stationary stepping test wherein the pace increases by 5 steps every 30 seconds using a metronome, lasting a maximum of 6 minutes. Clinical cardio-respiratory variables are simultaneously recorded. A portable metabolic analyzer, the Calibre Biometric Tracker, will be utilized to evaluate VO2 and VE (TV and RR). The Polar Sense of the Polar 10 heart rate monitor will measure HR on a continuous basis. The Train-Red Fyer NIRS Muscle Oxygen Sensor will be utilized to gather oxygenation data from muscle tissue.
  Interventions: Device: Portable mask for respiratory gas analysis
- Two day Cardio-Pulmonary Exercise Test (CPET) (Active Comparator): Prior to the CPET, spirometry is executed to predict the Maximum Voluntary Ventilation (MVV) from the Forced Expiratory Volume in one second (FEV1).The test is performed on a bicycle. The protocol is customized for each patient to achieve a fatigue-limited exercise duration of 8 to12 minutes. The predicted peak wattage is calculated according to a formula and by taking into account the patient's clinical profile. Patients start at 0 watts per minute. The intensity is increased until exhaustion (incremental step protocol) or if the test needs to be stopped for safety reasons. Patients are connected to an electrocardiogram (ECG), oximeter and blood pressure cuff. A mouthpiece is used to collect information about gas exchange.
  Interventions: Device: Cardio-pulmonary exercise test

INTERVENTIONS:
Device: Portable mask for respiratory gas analysis — This is a portable mask, which is connected to the SplendoHealth app. The Polar sens 10 heartrate monitor and TrainRed NIRS device are also connected to this app. The three devices (mask, heartrate monitor and NIRS) are measuring respiratory gases, heart rate and muscle tissue oxygenation simultanuously and at the end of the 6 min step test, you get an individual cardiorespiratory fitness report.
  Other Names: SplendoHealth app
  Arms: Two day 6-Minute Incremental Step Test (6 MIST)
Device: Cardio-pulmonary exercise test — Golden standard for measuring PEM: the double cardio-pulmonary exercise test on a bike.
  Other Names: CPET
  Arms: Two day Cardio-Pulmonary Exercise Test (CPET)

SUMMARY:
This study aims to evaluate exercise capacity and identify causes of Post-Exertional Symptom Exacerbation (PESE) in individuals with Long COVID. The investigators will compare the effectiveness of the Two-Day 6-Minute Incremental Step Test (6MIST) and the Cardiopulmonary Exercise Test (CPET) in detecting PESE. Additionally, the investigators will assess metabolism, mitochondrial function, autonomic symptoms, psychological factors, and physical activity. Participants will complete both the Two-Day 6MIST and the Two-Day CPET, with a one-month gap between them. Each test is performed on two consecutive days to assess the delayed symptom response. The subjective symptoms of PESE will also be measured through questionnaires. To explore potential causes of PESE, the investigators will measure metabolism using indirect calorimetry, bioelectrical impedance analysis and food diaries, mitochondrial dysfunction with NIRS technology, autonomic symptoms using the COMPASS-31 questionnaire, psychological factors with questionnaires and physical activity levels using an activity tracker. This study will determine if the Two-Day Step Test (6MIST) is a feasible alternative to the two-day CPET for measuring PESE and will help uncover underlying mechanisms contributing to symptom exacerbation.

ELIGIBILITY:
Inclusion Criteria:

* ≥18 years old
* Long COVID patients following the World Health Organization (WHO) criteria: "the continuation or development of new symptoms 3 months after the initial SARS-CoV-2 infection, with these symptoms lasting for at least 2 months with no other explanation"
* Previously active as described in the WHO recommendations for physical activity (minimal 150 minutes/week of moderate intensity aerobic physical activity OR minimal 75 minutes of vigorous intensity activity/week OR an equivalent combination of moderate- and vigorous-intensity activity throughout the week)
* Patient suffers from PESE as defined by the DePaul Symptom Questionnaire PEM (Post-Exertional Malaise) subscale
* Able to understand and sign written informed consent in Dutch, French or English

Exclusion Criteria:

* Any pre-existing conditions or new medical diagnosis that can alternatively explain the current symptoms
* Being unable to perform a cycle ergometer test as decided upon by the medical study team members
* Suffering from Chronic Obstructive Pulmonary Disease (COPD) GOLD classification category 2,3 or 4 (by the Global Initiative for Chronic Obstructive Lung Disease)
* Allergies to medical adhesive bandages
* Skin conditions aggravated by sunlight including Porphyria
* Participation in other interventional trials
* Mitochondrial diseases
* Pregnancy
* Lactation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2025-03-20 (Actual); Primary Completion 2025-07-03 (Actual); Study Completion 2025-07-03 (Actual)

PRIMARY OUTCOMES:
Difference in oxygen uptake at peak (VO2 peak) between day 1 and day 2 measured with the CPET compared to measured with the Calibre device | From day 1 and day 2 of experimental session 1 to day 1 and day 2 of experimental session 2, one month apart (±10 days)
  The goal is to show that the Calibre device is a feasible alternative to the CPET.
Difference in Rate of Perceived Exertion (RPE) measured with the CPET compared to measured with the Calibre device | RPE will be measured during two experimental sessions, each with two days, one month apart. On day 1, RPE is recorded 15 minutes (±15 min) before and after the test. On day 2, RPE is measured 24 hours (±120 min) after test 1 and before test 2.]
  Rate of Perceived Exertion is measured with the Borg RPE Scale which is a subjective measurement instrument. The scores range from 6 to 20, in which 6 is equal to no exertion at all and 20 is maximal exertion.
Resting Energy Expenditure (kcal/kg/day), measured through Indirect Calorimetry (IC) | Baseline (measured once, during the first study visit)
  Measuring Resting Energy Expenditure as part of the Directed Acyclic Graph (DAG).
Total Energy Expenditure (TEE) in kcal/kg/day, measured through Indirect Calorimetry (IC) | Baseline (measured once during the first study visit)
  Measuring Total Energy Expenditure as part of the DAG.
Phase angle (degrees), measured through Bioelectrical Impedance Analysis (BIA) | Baseline (measured once during the first study visit)
  Measuring Phase Angle as part of the DAG.
Muscle mass (kg/m2), measured through Bioelectrical Impedance Analysis (BIA) | Baseline (measured once during the first study visit)
  Measuring muscle mass as part of the DAG.
Fat mass index (kg/m2), measured through Bioelectrical Impedance Analysis (BIA) | Baseline (measured once during the first study visit)
  Measuring fat mass index as part of the DAG.
Fat-free mass index (kg/m²), measured through Bioelectrical Impedance Analysis (BIA) | Baseline (measured once during the first study visit)
  Measuring fat free mass index as part of the DAG.
Fat to fat-free mass ratio, measured through bioelectrical impedance analysis (BIA) | Baseline (measured once during the first study visit)
  Measuring fat-free mass ratio as part of the DAG.
Hydration (%), measured through Bioelectrical Impedance Analysis (BIA) | Baseline (measured once during the first study visit)
  Measuring hydration as part of the DAG.
Ratio of calorie and protein intake to individual need, measured through food diaries | Between day 1 of study visit and day 1 of experimental session
  Adequacy of feeding: the ratio between intake of calories and proteins and the individual need.
  Record of all food and drinks consumed over a 3-day period as part of the DAG.
Mean daily intake of calories, fats, proteins, and carbohydrates, measured through food diaries | Between day 1 of study visit and day 1 of experimental session
  Mean daily intake: calories, fats, proteins, carbohydrates Record of all food and drinks consumed over a 3-day period.
Oxygen availability as the partial pressure of oxygen (mitoPO2) (mmHg), measured through Near-infrared spectroscopy (NIRS) | Baseline (measured once during the first study visit)
  Measuring oxygen availability as the partial pressure of oxygen as part of the DAG.
Kinesiophobia with the Tampa Scale for Kinesiophobia (TSK) | Baseline (measured once during the first study visit)
  The Tampa Scale for Kinesiophobia (TSK) consists of 17 statements, each scored from 1 to 4, with 1 being 'strongly disagree' and 4 being 'strongly agree.' Higher scores indicate greater kinesiophobia. Measuring kinesiophobia as part of the DAG.
Ability to bounce back after stressful events with the Brief Resilience Scale (BRS) Questionnaire | Baseline (measured once during the first study visit)
  The Brief Resilience Scale (BRS) consists of 6 statements, each scored from 1 to 4, with 1 being 'strongly disagree' and 4 being 'strongly agree.' Higher scores indicate greater resilience. Measuring resilience as part of the DAG.
Coping style with the Ways of Coping (WAYS) Questionnaire | Baseline (measured once during the first study visit)
  Sixty-six statements about a stressful situation that participants experienced in the past week, for which they need to give a score ranging from 0 to 3, with 0 being "does not apply" or "not used," and 3 being "used a great deal". Measuring coping style as part of the DAG.
Autonomic symptoms, measured with the COMPASS-31 questionnaire | Baseline (measured once during the first study visit)
  Measuring autonomic symptoms as part of the DAG.
Level of Physical Activity (PA) and sedentary behavior assessed by accelerometry (activity tracker) | During 7 days before the first experimental session
  Using an actigraph, with a frequenncy of 60 Hertz, that participants wear at their hip on their dominant side. Measuring physical activity as part of the DAG.

SECONDARY OUTCOMES:
Change from Day 1 to Day 2 in Oxygen Uptake at First Ventilatory Threshold (VO₂ in ml/min/kg) during experimental session 1 or 2 (CPET) | From Day 1 to Day 2 during experimental session 1 or 2 (CPET)
Change from Day 1 to Day 2 in Oxygen uptake at peak (VO2 in ml/min/kg) during experimental session 1 and 2 (CPET & 6MIST)) | From Day 1 to Day 2 during experimental sessions 1 and 2 (CPET & 6MIST)
Change from Day 1 to Day 2 in Workload (Watts) at first ventilatory threshold during experimental session 1 or 2 (CPET) | From Day 1 to Day 2 during experimental session 1 or 2 (CPET)
Change from Day 1 to Day 2 in Workload (Watts) at peak during experimental session 1 or 2 (CPET) | From Day 1 to Day 2 during experimental session 1 or 2 (CPET)
Change from Day 1 to Day 2 in Heart Rate (bpm) peak during experimental sessions 1 and 2 (CPET & 6MIST)) | From Day 1 to Day 2 during experimental sessions 1 and 2 (CPET & 6MIST)
Change from Day 1 to Day 2 in Ventilation (VE) (Tidal Volume (TV) and Respiration Rate (RR)) during experimental sessions 1 and 2 (CPET 1 6MIST) | From Day 1 to Day 2 during experimental sessions 1 and 2 (CPET & 6MIST
Change from Day 1 to Day 2 in VE/VO2 slope during experimental sessions 1 and 2 (CPET and 6 MIST) | From Day 1 to Day 2 during experimental sessions 1 and 2 (CPET & 6MIST
Change from Day 1 to Day 2 in VO2/HR slope (= O2 pulse) during experimental sessions 1 and 2 (CPET and 6 MIST) | From Day 1 to Day 2 during experimental sessions 1 and 2 (CPET & 6MIST
Change from Day 1 to Day 2 in Respiratory Exchange Ratio (RER) = VCO2/VO2 during experimental sessions 1 or 2 (CPET) | From Day 1 to Day 2 during experimental session 1 or 2 (CPET)
Change from Day 1 to Day 2 in Cardiorespiratory Optimal Point (COP) = VO2/VE during experimental session 1 or 2 (CPET) | From Day 1 to Day 2 during experimental session 1 or 2 (CPET)

OTHER OUTCOMES:
Vaccination status of the participant | Baseline (inquired during the first study visit)
  Is the participant vaccinated or not, and with which vaccine.
Date of birth of the participant | Baseline (inquired during the first study visit)
  Date of birth of the participant. This is needed to make sure the participant is older than 18.
Ethnicity of the participant | Baseline (inquired during the first study visit)
  What is the ethnicity of the participant. (White, Hispanic/Latino, Black/African/African American, Asian, Native American/Indigenous)
BMI (kg/m²) | Baseline (calculated during the first study visit)
Hospitalization for COVID-19 | Baseline (inquired during the first study visit)
  Has the participant been hospitalized for his or her COVID infection, yes or no.
  If yes, has the participant been hospitalized in the ICU or not.
Educational level of the participant | Baseline (inquired during the first study visit)
  The highest degree of the participant.
Employement status of the participant | Baseline (inquired during the first study visit)
  The current employment status of the participant (employed full time or part-time, unemployed looking for work, unemployed not looking for work, self-employed, unable to work, student, retired).
Native language of the participant | Baseline (inquired during the first study visit)
  Native language of the participant (Dutch, French, English, German, Arabic, Other)

CONTACTS AND LOCATIONS:
Overall Officials: Elisabeth De Waele, MD, PhD, Principal Investigator — Universitair Ziekenhuis Brussel
Locations (2):
- Belgium (2):
  - Universitair Ziekenhuis Brussel, Jette, Brussels Capital
  - Universitair Ziekenhuis Brussel, Brussels, Jette

IPD SHARING:
Plan to Share IPD: No